CLINICAL TRIAL: NCT04438863
Title: A Descriptive Pilot Study of Daily Home Spirometry for Early Detection of Pulmonary Complications in High Risk Patients With COVID19
Brief Title: Daily Home Spirometry for Early Detection of Pulmonary Complications in Patients With COVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Liran Levy, Transplant pulmonologist, Sheba Medical Center
Other Study IDs: SHEBA-20-7022-SMC-LL-CTIL
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: home spirometry — portable hand-held spirometer to collect and store daily spirometric data (including FVC, FEV1, forced expiratory flow after 25 to 75% of vital capacity has been expelled, and peak flow).

SUMMARY:
The aim of this preliminary study is to describe the potential decline in forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) as measured by home spirometry in high-risk subjects infected with COVID-19. We hypothesize that the magnitude of such a decline in FEV1 and/or FVC may be associated with clinical deterioration and hospitalization. The study will ultimately inform a larger subsequent RCT that will evaluate the efficacy of home spirometry in the early detection (pre respiratory symptoms) of respiratory complications and therefore prompt early medical attention which is a key for improving outcome.

ELIGIBILITY:
Inclusion Criteria:

1. without dyspnea and with no evidence of pneumonia, ARDS, organ failure or requiring admission to ICU.
2. All patients ≥55 years age or ≥1 risk factor for disease complications (prior pulmonary, kidney or cardiovascular disease, diabetes mellitus, hypertension, bone merrow suppression, solid organ transplant, HIV with CD4<250, heavy smoker, BMI >30). All participants will sign a written informed consent.

Exclusion Criteria:

1. Patients unable to perform spirometry
2. contraindications for spirometry (hemoptysis, active tuberculosis, syncope associated with forced exhalation or increased risk for spirometry)
3. adhere to the follow-up protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: confirmed COVID19 patients (hospitalized or not hospitalized) with mild to moderate symptoms.
  (low grade fever, cough, anosmia, fatigue, discomfort, anorexia or other gastrointestinal symptoms)
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-08-08 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | number of participants hospitalized in a time frame of a year
  participants that are hospitalized

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No